CLINICAL TRIAL: NCT01370447
Title: Emergency Use Protocol for EPI-743 in Acutely Ill Patients With Inherited Mitochondrial Respiratory Chain Disease Within 90 Days of End-of-Life Care
Brief Title: EPI-743 for Mitochondrial Respiratory Chain Diseases
Status: No longer available | Type: Expanded Access
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: EPI-2009-1
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Mitochondrial Diseases
Keywords: Leigh syndrome; MELAS; Kearns-Sayre; Alper's; Inherited mitochondrial disease; Friedreich's ataxia; POLG1 deficiency
MeSH Terms: conditions — Mitochondrial Diseases; Leigh Disease; MELAS Syndrome; Friedreich Ataxia | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: EPI-743 — EPI-743 (oral solution [100 mg/mL] or liquid-filled capsules [100 mg or 200 mg]) will be administered per dose and schedule specified in the arm.
  Other Names: Vincerinone, Vatiquinone

SUMMARY:
This study will evaluate the safety and efficacy of EPI-743 in participants with severe mitochondrial respiratory chain diseases who are considered to be within 90 days of end-of-life care.

ELIGIBILITY:
Inclusion criteria:

1. Participants with genetic diagnosis: Genetically confirmed diagnosis of Inherited mitochondrial respiratory chain disease
2. Participants with clinical diagnosis: Diagnosis of inherited mitochondrial disease absent genetic confirmation; Specifically, participants must meet the diagnostic criteria of "definite" or "probable" mitochondrial disease as defined by Bernier et al., 2002
3. Deemed by principal investigator to be within 90 days of end-of-life hospice/terminal care
4. Male or female age > one year
5. Hematocrit within normal range for age group
6. Agreement to use contraception if within reproductive years
7. Participant or participant's guardian able to consent and comply with protocol requirements
8. Presence of caregiver to ensure study compliance
9. Abstention from use of all pill-form dietary supplements and non-prescribed medications (except as allowed by the investigator)
10. Abstention from foods or beverages or bars fortified with Coenzyme Q10, vitamin E, super-fortified "functional" foods or beverages
11. Abstention from use of idebenone
12. Clinically staged with a Mitochondrial Disease Scale such as the Newcastle Score

Exclusion criteria:

1. Allergy to EPI-743, vitamin E or sesame oil
2. Clinical history of bleeding or abnormal prothrombin time (PT)/partial thromboplastin time (PTT) (excluding anticoagulation Rx)
3. Hepatic insufficiency with liver function tests (LFTs) greater than two times normal
4. Renal insufficiency requiring dialysis
5. Fat malabsorption syndromes precluding drug absorption
6. Any other concurrent inborn errors of metabolism
7. Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis
8. Pregnancy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Enns, MB, ChB, Principal Investigator — Stanford University
Locations (16):
- United States (16):
  - UCLA, Los Angeles, California
  - CHOC Children's Clinic, Orange, California
  - Lucille Packard Children's Hospital, Palo Alto, California
  - UCSD, San Diego, California
  - Stanford Children's Health, Stanford, California
  - Emory University, Decatur, Georgia
  - CUMC (Columbia University), New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - MUSC, North Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - UTH, Houston, Texas
  - Naval Hospital, Bremerton, Bremerton, Washington
  - Seattle Children's Hospital, Seattle, Washington